CLINICAL TRIAL: NCT00567112
Title: An Open-Label, Randomized, Partially Fixed-Sequence, 4-Period Crossover Study to Assess the Pharmacokinetics After Administration of the DFC and OCT Formulations and the Food Effect on the OCT Formulation of MK-0941 in Patients With Type 2 Diabetes
Brief Title: Study to Evaluate the Pharmacokinetics & Food Effect of MK-0941 in Adults With Type 2 Diabetes (MK-0941-009)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0941-009; 2007_652 (Other: Merck Registration ID); MK-0941-009 (Other: Merck Protocol ID)
Record Dates: First submitted 2007-11-30; First posted 2007-12-04 (Estimated); Results first posted 2012-09-05 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Postprandial Period

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- DFC (fasted) (Experimental)
  Interventions: Drug: 10 mg MK-0941 DFC (fasted)
- OCT (fasted) (Experimental)
  Interventions: Drug: 10 mg MK-0941 OCT (fasted)
- OCT (after meal) (Experimental)
  Interventions: Drug: 10 mg MK-0941 OCT (after meal)
- OCT (before meal) (Active Comparator)
  Interventions: Drug: 10 mg MK-0941 OCT (before meal)

INTERVENTIONS:
Drug: 10 mg MK-0941 DFC (fasted) — single dose of 10 mg MK-0941 dry filled capsules (DFC) administered in a fasted state
  Arms: DFC (fasted)
Drug: 10 mg MK-0941 OCT (after meal) — single dose of 10 mg MK-0941 oral compressed tablet (OCT) administered after consumption of a high-fat meal
  Arms: OCT (after meal)
Drug: 10 mg MK-0941 OCT (before meal) — single dose of 10 mg MK-0941 oral compressed tablet (OCT) administered before consumption of a standard breakfast
  Arms: OCT (before meal)
Drug: 10 mg MK-0941 OCT (fasted) — single dose of 10 mg MK-0941 oral compressed tablet (OCT) administered in a fasted state
  Arms: OCT (fasted)

SUMMARY:
A study to compare the pharmacokinetics (PK) of the dry filled capsule (DFC) & oral compressed tablet (OCT) formulations of MK-0941-009 & to assess the effect of food on the OCT formulation.

ELIGIBILITY:
Inclusion Criteria:

* Males or females (of non-childbearing potential) between the ages of 18 to 70
* Participants have been diagnosed with Type 2 Diabetes
* Participants are nonsmokers for at least 6 months

Exclusion Criteria:

* Participant should not be diagnosed with Type 1 diabetes
* Participant should not be receiving insulin or PPAR gamma agonists for 12 weeks prior to study start
* Participant has a recent history of eye infection or other inflammatory eye condition within 2 weeks prior to study start
* Participant has been diagnosed with glaucoma or is blind
* Participant has had trauma to one or both eyes
* Participant has had major surgery, donated blood or participated in another clinical study in the past 4 weeks
* Participant is a regular user of illicit drugs or has a history of drug, including alcohol, abuse in the past 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-11; Primary Completion 2008-02 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group ABCD: * Period 1: Dry Filled Capsule (DFC) (fasted)
  * Period 2: Oral Compressed Tablet (OCT) (fasted)
  * Period 3: OCT (after meal)
  * Period 4: OCT (before meal)
- Treatment Group BACD: * Period 1: OCT (fasted)
  * Period 2: DFC (fasted)
  * Period 3: OCT (after meal)
  * Period 4: OCT (before meal)
- Treatment Group BCD: * Period 1: Not Applicable
  * Period 2: OCT (fasted)
  * Period 3: OCT (after meal)
  * Period 4: OCT (before meal)
Period: Treatment Period 1 (3 Days)
Arm/Group | Treatment Group ABCD | Treatment Group BACD | Treatment Group BCD
Started | 7 | 8 | 0
Completed | 7 | 8 | 0
Not Completed | 0 | 0 | 0
Period: Washout Period 1 (3 Days)
Arm/Group | Treatment Group ABCD | Treatment Group BACD | Treatment Group BCD
Started | 7 | 8 | 0
Completed | 7 | 8 | 0
Not Completed | 0 | 0 | 0
Period: Treatment Period 2 (3 Days)
Arm/Group | Treatment Group ABCD | Treatment Group BACD | Treatment Group BCD
Started | 7 | 8 | 3 (3 new participants added to Treatment Group ABCD & received treatment sequence BCD for Periods 2-4)
Completed | 7 | 7 | 3
Not Completed | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Period: Washout Period 2 (3 Days)
Arm/Group | Treatment Group ABCD | Treatment Group BACD | Treatment Group BCD
Started | 7 | 7 | 3
Completed | 7 | 7 | 3
Not Completed | 0 | 0 | 0
Period: Treatment Period 3 (3 Days)
Arm/Group | Treatment Group ABCD | Treatment Group BACD | Treatment Group BCD
Started | 7 | 7 | 3
Completed | 7 | 7 | 3
Not Completed | 0 | 0 | 0
Period: Washout Period 3 (3 Days)
Arm/Group | Treatment Group ABCD | Treatment Group BACD | Treatment Group BCD
Started | 7 | 7 | 3
Completed | 4 | 7 | 3
Not Completed | 3 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Period: Treatment Period 4 (3 Days)
Arm/Group | Treatment Group ABCD | Treatment Group BACD | Treatment Group BCD
Started | 4 | 7 | 3
Completed | 4 | 7 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Randomized: Includes the 15 participants who were randomized and started the study in Treatment Period 1 (Baseline) and the 3 additional participants who were subsequently randomized and started the study in Treatment Period 2.
Arm/Group | All Randomized
Number analyzed (Participants) | 18
Age, Customized [Number; unit: participants]
  ≥ 35 and ≤ 69 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC)(0-∞) for Oral Compressed Tablet (OCT) (Fasted) and Dry Filled Capsule (DFC) (Fasted)
Time Frame: From study drug administration to 72 hours post-administration
Population: Participants with AUC(0-∞) measurements
Measure: Least Squares Mean (Full Range); unit: nM*hr
Groups:
- OCT (Fasted): Participants receiving a single dose of 10 mg MK-0941 OCT administered in a fasted state
- DFC (Fasted): Participants receiving a single dose of 10 mg MK-0941 DFC administered in a fasted state
Arm/Group | OCT (Fasted) | DFC (Fasted)
Number analyzed (Participants) | 18 | 14
nM*hr | 763.76 [579.52 to 1681.47] | 776.41 [470.04 to 1698.00]
Statistical Analysis 1: Comparison: OCT (Fasted) vs DFC (Fasted); OCT (fasted)/DFC (fasted); Test type: Non-Inferiority or Equivalence — Geometric Mean Ratio of OCT (fasted)/DFC (fasted); p > 0.200, ANOVA; Geometric Mean Ratio = 0.98, 90% CI 2-sided [0.92 to 1.05]

2. Primary Outcome: Maximum Concentration (Cmax) for OCT (Fasted) and DFC (Fasted)
Time Frame: From study drug administration to 72 hours post-administration
Population: Participants with Cmax measurements
Measure: Least Squares Mean (Full Range); unit: nM
Arm/Group | OCT (Fasted) | DFC (Fasted)
Number analyzed (Participants) | 18 | 15
nM | 241.37 [96.84 to 607.42] | 246.92 [78.17 to 539.93]
Statistical Analysis 1: Comparison: OCT (Fasted) vs DFC (Fasted); OCT (fasted)/DFC (fasted); Test type: Non-Inferiority or Equivalence — Geometric Mean Ratio of OCT (fasted)/DFC (fasted); p > 0.200, ANOVA; Geometric Mean Ratio = 0.98, 90% CI 2-sided [0.80 to 1.19]

3. Secondary Outcome: AUC(0-∞) for OCT (Fasted) and OCT (After Meal)
Time Frame: From study drug administration to 72 hours post-administration
Population: Participants with AUC(0-∞) measurements
Measure: Least Squares Mean (Full Range); unit: nM*hr
Groups:
- OCT (After Meal): Participants receiving a single dose of 10 mg MK-0941 OCT administered after consumption of a high-fat meal
Arm/Group | OCT (Fasted) | OCT (After Meal)
Number analyzed (Participants) | 18 | 17
nM*hr | 763.76 [579.52 to 1681.47] | 702.08 [467.62 to 1375.86]
Statistical Analysis 1: Comparison: OCT (Fasted) vs OCT (After Meal); OCT (after meal)/OCT (fasted); Test type: Non-Inferiority or Equivalence — Geometric Mean Ratio of OCT (after meal)/OCT (fasted); p = 0.026, ANOVA; Geometric Mean Ratio = 0.92, 90% CI 2-sided [0.86 to 0.98]

4. Secondary Outcome: Cmax of OCT (Fasted) and OCT (After Meal)
Time Frame: From study drug administration to 72 hours post-administration
Population: Participants with Cmax measurements
Measure: Least Squares Mean (Full Range); unit: nM
Arm/Group | OCT (Fasted) | OCT (After Meal)
Number analyzed (Participants) | 18 | 17
nM | 241.37 [96.84 to 607.42] | 143.51 [64.13 to 268.08]
Statistical Analysis 1: Comparison: OCT (Fasted) vs OCT (After Meal); OCT (after meal)/OCT (fasted); Test type: Non-Inferiority or Equivalence — Geometric Mean Ratio OCT (after meal)/OCT (fasted); p < 0.001, ANOVA; Geometric Mean Ratio = 0.59, 90% CI 2-sided [0.49 to 0.72]

5. Primary Outcome: Time to Reach Cmax (Tmax) for OCT (Fasted) and DFC (Fasted)
Time Frame: From study drug administration to 72 hours post-administration
Population: Participants with Tmax measurements
Measure: Median (Full Range); unit: hours
Arm/Group | OCT (Fasted) | DFC (Fasted)
Number analyzed (Participants) | 18 | 15
hours | 1.00 [0.50 to 4.00] | 1.00 [0.20 to 1.50]
Statistical Analysis 1: Comparison: OCT (Fasted) vs DFC (Fasted); OCT (fasted)/DFC (fasted); Test type: Superiority or Other; p > 0.200, ANOVA

6. Primary Outcome: Half Life (t½) for OCT (Fasted) and DFC (Fasted)
Time Frame: From study drug administration to 72 hours post-administration
Population: Participants with t1/2 measurements
Measure: Median (Full Range); unit: hours
Arm/Group | OCT (Fasted) | DFC (Fasted)
Number analyzed (Participants) | 18 | 14
hours | 9.85 [3.90 to 27.00] | 8.05 [5.30 to 38.40]
Statistical Analysis 1: Comparison: OCT (Fasted) vs DFC (Fasted); OCT (fasted)/DFC (fasted); Test type: Superiority or Other; p > 0.200, ANOVA

7. Secondary Outcome: Tmax for OCT (Fasted) and OCT (After Meal)
Time Frame: From study drug administration to 72 hours post-administration
Population: Participants with Tmax measurements
Measure: Median (Full Range); unit: hours
Arm/Group | OCT (Fasted) | OCT (After Meal)
Number analyzed (Participants) | 18 | 17
hours | 1.00 [0.50 to 4.00] | 2.00 [1.00 to 4.00]
Statistical Analysis 1: Comparison: OCT (Fasted) vs OCT (After Meal); OCT (after meal)/OCT (fasted); Test type: Superiority or Other; p < 0.001, ANOVA

8. Secondary Outcome: t1/2 for OCT (Fasted) and OCT (After Meal)
Time Frame: From study drug administration to 72 hours post-administration
Population: Participants with t1/2 measurements
Measure: Median (Full Range); unit: hours
Arm/Group | OCT (Fasted) | OCT (After Meal)
Number analyzed (Participants) | 18 | 17
hours | 9.85 [3.90 to 27.00] | 9.60 [3.30 to 23.20]
Statistical Analysis 1: Comparison: OCT (Fasted) vs OCT (After Meal); OCT (after meal)/OCT (fasted); Test type: Superiority or Other; p > 0.200, ANOVA

ADVERSE EVENTS:
Time Frame: From first dose of study drug administration through to 72 hours post-administration
Groups:
- OCT (Before Meal): Participants receiving a single dose of 10 mg MK-0941 OCT administered before consumption of a standard breakfast
Arm/Group | OCT (Fasted) | OCT (After Meal) | OCT (Before Meal) | DFC (Fasted)
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17 | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 6/18 | 7/17 | 3/14 | 4/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OCT (Fasted) (N=18) | OCT (After Meal) (N=17) | OCT (Before Meal) (N=14) | DFC (Fasted) (N=15)
Asthenia (General disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Catheter site pain (General disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 1
Infusion site erythema (General disorders) | 1 | 2 | 0 | 0
Infusion site pain (General disorders) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Tongue Blistering (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.